CLINICAL TRIAL: NCT07374718
Title: Optimization and Verification of Quality Control Indicators for Coronary Revascularization Based on Antiplatelet Therapy: Safety and Efficacy of De-escalation Dual Antiplatelet Therapy in Moderate-to-high Ischemic Risk and High Bleeding Risk ACS Patients After BioFreedom™ Drug-Coated Coronary Stenting
Brief Title: Safety and Efficacy of De-escalation Dual Antiplatelet Therapy After BioFreedom™ Stenting in ACS Patients With Moderate-to-high Ischemic and High Bleeding Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Director, clinical professor, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZD0546702-RCT
Record Dates: First submitted 2026-01-20; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-09

CONDITIONS: Acute Coronary Syndrome (ACS); High Bleeding Risk(HBR); Coronary Artery Disease (CAD)
Keywords: Dual Antiplatelet Therapy (DAPT); Acute Coronary Syndrome (ACS); High Bleeding Risk (HBR); Percutaneous Coronary Intervention (PCI); Quality Control Indicators; Coronary Revascularization; Real-World Research; Bleeding Events; Ischemic Events; Post-PCI Prognosis
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Interventional Model Description This study is a parallel-group RCT aiming to assess the safety and efficacy of IVUS-guided BioFreedom™ stenting plus 1-month DAPT de-escalation versus angiography-guided conventional DES stenting plus 12-month DAPT in ACS patients with moderate-to-high ischemic and high bleeding risk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular ultrasound (IVUS)-guided implantation of BioFreedom™ drug-coated coronary stent system (Experimental): 1 month of dual antiplatelet therapy (DAPT: aspirin 100mg/day + clopidogrel 75mg/day or ticagrelor 90mg twice daily) followed by 11 months of single antiplatelet therapy (SAPT: clopidogrel 75mg/day or ticagrelor 90mg twice daily)
  Interventions: Device: IVUS-guided BioFreedomTM Drug-Coated Stent Implantation + 1-Month DAPT Followed by 11-Month P2Y12 Inhibitor Monotherapy
- Angiography-guided implantation of other drug-eluting stents (DES) (Other): 12 months of conventional dual antiplatelet therapy (DAPT: aspirin 100mg/day + clopidogrel 75mg/day or ticagrelor 90mg twice daily)
  Interventions: Device: Angiography-guided Conventional Drug-Eluting Stent Implantation + 12-Month Dual Antiplatelet Therapy (Aspirin + P2Y12 Inhibitor)

INTERVENTIONS:
Device: IVUS-guided BioFreedomTM Drug-Coated Stent Implantation + 1-Month DAPT Followed by 11-Month P2Y12 Inhibitor Monotherapy — Intravascular ultrasound (IVUS)-guided implantation of BioFreedom™ polymer-free drug-coated stent, followed by 1-month dual antiplatelet therapy (DAPT: aspirin + P2Y12 inhibitor) and 11-month P2Y12 inhibitor monotherapy for ACS patients with high bleeding and intermediate-to-high ischemic risk.
  Arms: Intravascular ultrasound (IVUS)-guided implantation of BioFreedom™ drug-coated coronary stent system
Device: Angiography-guided Conventional Drug-Eluting Stent Implantation + 12-Month Dual Antiplatelet Therapy (Aspirin + P2Y12 Inhibitor) — Coronary angiography-guided implantation of conventional drug-eluting stent (DES), with 12-month standard DAPT (aspirin + P2Y12 inhibitor) for the same patient population.
  Arms: Angiography-guided implantation of other drug-eluting stents (DES)

SUMMARY:
Patients with acute coronary syndrome (ACS) who have both high ischemic risk and high bleeding risk represent a challenging population following percutaneous coronary intervention (PCI), as prolonged dual antiplatelet therapy (DAPT) may reduce ischemic events but increases bleeding complications.This prospective, multicenter, randomized controlled study evaluates the safety and effectiveness of an optimized PCI and antiplatelet therapy strategy in ACS patients with moderate-to-high ischemic risk and high bleeding risk. Eligible patients will be randomized in a 1:1 ratio to either an experimental strategy consisting of intravascular ultrasound-guided implantation of a polymer-free drug-coated stent followed by one month of DAPT and subsequent single antiplatelet therapy, or a control strategy consisting of angiography-guided implantation of contemporary drug-eluting stents followed by standard 12-month DAPT.The primary hypothesis is that the experimental strategy will reduce the incidence of net adverse clinical events, defined as a composite of ischemic and bleeding outcomes, compared with conventional PCI and prolonged DAPT. Participants will be followed for 12 months after the index procedure.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled trial designed to evaluate an optimized revascularization and antiplatelet therapy strategy in patients with acute coronary syndrome (ACS) who present with both moderate-to-high ischemic risk and high bleeding risk.Eligible patients aged 18 years or older who meet Academic Research Consortium-High Bleeding Risk criteria and have an OPT-CAD score of 90 or higher will be randomized in a 1:1 ratio to an experimental group or a control group. Patients in the experimental group will undergo intravascular ultrasound-guided PCI with implantation of a polymer-free drug-coated coronary stent, followed by one month of dual antiplatelet therapy consisting of aspirin and a P2Y12 inhibitor, and subsequent single antiplatelet therapy. Patients in the control group will undergo angiography-guided PCI with implantation of contemporary drug-eluting stents and receive standard dual antiplatelet therapy for 12 months.Clinical follow-up will be conducted at discharge and at 30 days, 6 months, and 12 months after the index procedure. Clinical data collected during follow-up will include ischemic events, bleeding events, antiplatelet therapy use, and adverse events.The primary endpoint is the incidence of net adverse clinical events at 12 months, defined as a composite of ischemic and bleeding outcomes, including cardiac death, myocardial infarction, ischemic stroke, definite stent thrombosis, clinically driven target vessel revascularization, or bleeding events classified according to the Bleeding Academic Research Consortium criteria. Secondary endpoints include clinically relevant bleeding and ischemic outcomes.Study data will be collected using a centralized electronic data capture system with predefined data validation rules and audit trails. Data quality will be ensured through investigator training, standardized operating procedures, automated range and consistency checks, and regular site monitoring with source data verification against source documents. A predefined data dictionary will describe all registry variables, including definitions, coding information, and clinically relevant ranges where applicable. Missing data will be addressed according to a prespecified statistical analysis plan.The planned sample size is 468 participants, providing adequate statistical power to detect differences in the primary endpoint using an intention-to-treat analytical approach.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* ACS patients with high bleeding risk (meeting the ARC-HBR criteria)
* Moderate-to-high ischemic risk (OPT-CAD score ≥ 90)
* Predicted by the investigator to be able to tolerate 12 months of DAPT
* Voluntarily participate and sign the informed consent form, and be willing to receive the designated follow-up of this trial at specific time points
* Coronary artery lesions are primary and in-situ coronary artery lesions
* Target lesion diameter stenosis ≥ 70% or ≥ 50% (visual estimation) accompanied by evidence of myocardial ischemia

Exclusion Criteria:

* Patients with known allergy or contraindication to P2Y12 inhibitors, aspirin, or contrast agents
* Patients planning to undergo surgical intervention within 12 months
* Left Ventricular Ejection Fraction (LVEF) < 35%
* Patients with contraindications to PCI
* Patients with a history of substance abuse (alcohol, cocaine, heroin, etc.), or with an expected life expectancy of less than 1 year
* Subjects with poor compliance or judged by the investigator to be unsuitable for participating in the study
* Female patients who are planning to be pregnant or are pregnant/lactating, and male patients planning to impregnate
* Chronic total occlusion lesions
* Lesions involving the left main coronary artery
* Severe calcified and tortuous lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
The 12-month incidence of Net Adverse Clinical Events (NACE) | 12 Months
  NACE is defined as a composite endpoint of bleeding and ischemic events, including cardiac death, myocardial infarction, ischemic stroke, definite stent thrombosis, clinically driven target vessel revascularization, or any bleeding (BARC defined type 1, 2, 3, 5 bleeding according to the Bleeding Academic Research Consortium [BARC]) (for superiority assessment).

SECONDARY OUTCOMES:
The 12-month incidence of clinically relevant bleeding events (for superiority assessment) | 12 Months
Clinically relevant bleeding events refer to BARC defined type 2, 3, 5 bleeding | 12 Months
The incidence of NACE and clinically relevant bleeding events (including BARC type 2, 3, 5 bleeding) at 30 days and 6 months | 30 days and 6 months
Incidence of clinically driven target lesion revascularization (CD-TLR)at 30 days, 6 months, and 12 months | 30 days, 6 months, and 12 months
Incidence of major bleeding events (including BARC type 3, 5 bleeding)at 30 days, 6 months, and 12 months | 30 days, 6 months, and 12 months
Incidence of BARC type 1, 2, 3, 5 bleeding at 30 days, 6 months, and 12 months | 30 days, 6 months, and 12 months
Incidence of definite or probable in-stent thrombosis events at 30 days, 6 months, and 12 months | 30 days, 6 months, and 12 months
  Thrombotic events refer to definite or probable in-stent thrombosis as defined by the Academic Research Consortium (ARC).
Incidence of Target Vessel Failure (TVF) | 30 days, 6 months, and 12 months
  Defined as a composite endpoint of cardiac death, target vessel myocardial infarction, and clinically driven target vessel revascularization.
Incidence of Major Adverse Cardiovascular Events (MACE) | 30 days, 6 months, and 12 months
  Defined as a composite endpoint of cardiac death, myocardial infarction, and target vessel revascularization.
Incidence of Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 30 days, 6 months, and 12 months
  Defined as a composite endpoint of all-cause death, myocardial infarction, stroke, or clinically driven coronary revascularization.
Incidence of all-cause death | 30 days, 6 months, and 12 months
Incidence of cardiac death | 30 days, 6 months, and 12 months
Incidence of ischemic stroke | 30 days, 6 months, and 12 months
Incidence of target vessel revascularization | 30 days, 6 months, and 12 months
DAPT discontinuation rate | 30 days, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tan Mengqin, Yin Chune, Wang Fujun. Interpretation of the 2018 Updated Universal Definition of Myocardial Infarction. Journal of Practical Electrocardiology 2018; 27(06): 381-5.
- [Background] Cao D, Vranckx P, Valgimigli M, et al. One- versus three-month dual antiplatelet therapy in high bleeding risk patients undergoing percutaneous coronary intervention for non-ST-segment elevation acute coronary syndromes. EuroIntervention 2024; 20(10): e630-e42.
- [Background] Valgimigli M, Frigoli E, Heg D, et al. Dual antiplatelet therapy after PCI in patients at high bleeding risk. New England Journal of Medicine 2021; 385(18): 1643-55.
- [Background] Urban P, Meredith IT, Abizaid A, et al. Polymer-free drug-coated coronary stents in patients at high bleeding risk. New England Journal of Medicine 2015; 373(21): 2038-47.
- [Background] Byrne RA, Rossello X, Coughlan JJ, et al. 2023 ESC Guidelines for the management of acute coronary syndromes: Developed by the task force on the management of acute coronary syndromes of the European Society of Cardiology (ESC). European Heart Journal: Acute Cardiovascular Care 2024; 13(1): 55-161.
- [Background] Rao SV, O'Donoghue ML, Ruel M, et al. 2025 ACC/AHA/ACEP/NAEMSP/SCAI Guideline for the Management of Patients With Acute Coronary Syndromes: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation 2025.
- [Background] Chinese Society of Cardiology, Editorial Board of Chinese Journal of Cardiology. Guidelines for the Diagnosis and Treatment of Non-ST-segment Elevation Acute Coronary Syndrome (2024). Chinese Journal of Cardiology 2024; 52(06): 615-46.
- [Background] Liu Mingbo, He Xinye, Yang Xiaohong, Wang Zengwu, Hu Shengshou. Summary of "China Cardiovascular Health and Disease Report 2023" (Epidemiology of Cardiovascular Diseases and Status of Interventional Diagnosis and Treatment). Chinese Journal of Interventional Cardiology 2024; 32(10): 541-50.
- [Background] Yin Peng, Qi Jinlei, Liu Yunning, et al. China's Disease Burden Study Report 2005-2017. Chinese Circulation Journal 2019; 34(12): 1145-54.
- [Background] Li Pengxiao. Long-term Prognosis and Influencing Factors of ACS Patients with High Bleeding Risk after PCI [Master's Thesis]; 2023.
- [Background] Ge Z, Kan J, Gao X, et al. Ticagrelor alone versus ticagrelor plus aspirin from month 1 to month 12 after percutaneous coronary intervention in patients with acute coronary syndromes (ULTIMATE-DAPT): a randomised, placebo-controlled, double-blind clinical trial. The Lancet 2024; 403(10439): 1866-78.
- [Background] Li X, Ge Z, Kan J, et al. Intravascular ultrasound-guided versus angiography-guided percutaneous coronary intervention in acute coronary syndromes (IVUS-ACS): a two-stage, multicentre, randomised trial. The Lancet 2024; 403(10439): 1855-65.
- [Background] Valgimigli M, Frigoli E, Heg D, et al. Dual Antiplatelet Therapy after PCI in Patients at High Bleeding Risk. New England Journal of Medicine 2021; 385(18): 1643-55.